CLINICAL TRIAL: NCT00892840
Title: Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-820836 in Healthy Subjects
Brief Title: Multiple-Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN162-002; 2008-008488-86
Record Dates: First submitted 2009-05-02; First posted 2009-05-05 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — 6-(2-methyl-4-(2-naphthyl)-1,2,3,4-tetrahydroisoquinolin-7-yl)pyridazin-3-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panels 1 to 7 (BMS-820836 or Placebo) (Experimental)
  Interventions: Drug: BMS-820836; Drug: Placebo

INTERVENTIONS:
Drug: BMS-820836 — Oral Solution, Oral, 0.1 mg to 4 mg, Once daily, 14 days
Drug: Placebo — Oral Solution, Oral, 0 mg, Once daily, 14 days

SUMMARY:
The purpose of this study is to determine the safety and tolerability of BMS-820836 after multiple doses

ELIGIBILITY:
Inclusion Criteria:

* Panels 1-6: Healthy Male Subjects
* Panel 7: Females
* Ages 21 to 55, inclusive
* Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* Any major surgery within 4 weeks of study drug administration
* History of cholecystectomy
* History of glaucoma or a confirmed intraocular pressure indicative of glaucoma at screening. (Normal IOP <21 mmHg)
* Confirmed QTc (Fridericia) value ≥ 450 msec
* Confirmed QT ≥ 500 msec
* Confirmed PR ≥ 210 msec
* Confirmed QRS ≥ 120 msec
* Confirmed resting supine systolic blood pressure > 140 mmHg
* Confirmed resting supine diastolic blood pressure > 90 mmHg
* Confirmed resting heart rate < 45 bpm or > 100 bpm
* Orthostatic vital sign changes (ie., a decrease in systolic blood pressure from supine to standing > 40 mmHg and an increase in heart rate from supine to standing > 20 bpm) or symptoms of orthostasis
* History of peppermint allergies
* Exposure to any investigational drug or placebo within 12 weeks of study drug administration

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of BMS-820836 following multiple-dose administration | Within 27 days (+/- 2 days) of first dose

SECONDARY OUTCOMES:
To assess the pharmacodynamics of BMS-820836 | Within 27 days of first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Uppsala, Sweden

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx